CLINICAL TRIAL: NCT04544553
Title: To Understand the Barriers and Facilitators of Diabetic Retinopathy Screening & Follow-up: An Exploratory Study From India and Thailand
Brief Title: Barriers to Eye Screening for People With Diabetes in India
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lions Club International Foundation (Other)
Responsible Party: Principal Investigator, Rajiv Raman, Senior Consultant (Ophthalmologist), Sankara Nethralaya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 731-2018-P
Record Dates: First submitted 2020-09-03; First posted 2020-09-10 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Diabetic Macular Edema
Keywords: screening; follow-up; short message service

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMS reminder (Other): This arm receive SMS reminder for the follow-up of DR Screening
  Interventions: Other: SMS reminder
- No SMS reminder (Other): This arm did not receive SMS reminder for the follow-up of DR Screening
  Interventions: Other: No SMS reminder

INTERVENTIONS:
Other: SMS reminder — The group receives reminder for the follow-up at 1 week and 2 days prior to their scheduled appointments.
  Arms: SMS reminder
Other: No SMS reminder — The group did not receives any SMS regarding scheduled appoinments.
  Arms: No SMS reminder

SUMMARY:
Brief Summary: Diabetic retinopathy (DR) is a leading cause of visual impairment and has major public health implications globally and especially in countries such as India where the prevalence of diabetes is high. With timely screening and intervention, the disease progression to blindness can be prevented but several barriers exist to the provision of care. The long term aim is to identify the barriers to DR screening and to plan potential interventional strategies. From the qualitative study, the reasons such as lack of awareness or knowledge, distance to travel, lack of reminder system were identified as a reason for poor follow-up. This lead to the development of interventional strategies.

This was a randomized, investigator-masked clinical trial that was conducted in a tertiary eye care centre in South India. Consecutive patients with diabetes who were residents in Chennai and its vicinity of approximately 100 km radius and who were undergoing repeated intravitreal injections for DME were recruited into the trial. The aim of the study is to investigate the effect of SMS informational reminders among patients with Diabetic macular edema for the follow-up. They study consists of 2 groups, SMS reminder group receives the reminders 1 week and 2 days prior to the scheduled appointments with the concerned doctor on a particular date and time, whereas other group does not receive any reminders for the appointment schedule. After the follow-up, the patients will be screened for the attendance at the review visit.

ELIGIBILITY:
Inclusion Criteria:

* Adults with > 40 years of age
* Diagnosed as centre involving Diabetic macular edema (DME)
* Patients who received intravitreal injections for DME
* Ability to give informed consent

Exclusion Criteria:

* Patients from outside the area of residence who stayed more than 100 km from the hospital
* Patients with ocular co-morbidities other than DME

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2019-08-14 (Actual); Study Completion 2019-08-14 (Actual)

PRIMARY OUTCOMES:
Attendance rates in patients with diabetic macular edema receiving short messaging services | 7 months
  To investigate the effect of SMS informational reminders on adherence with scheduled eye examinations among patients with center involving DME receiving intravitreal injections in a tertiary eye care institute in South India.

CONTACTS AND LOCATIONS:
Locations (1):
- Rajiv Raman, Chennai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No
The datasets generated during and/or analysed during the study are not publicly available, as it against the organization hospital policy. But are available from the corresponding author on reasonable request.

REFERENCES:
- [Derived] Kumar G, Velu S, Prakash VJ, Kumar S, Sivaprasad S, Sharma A, Raman R. Attendance Rate in Patients with Diabetic Macular Edema Receiving Short Messages. Ophthalmol Retina. 2021 Oct;5(10):1054-1056. doi: 10.1016/j.oret.2021.03.005. Epub 2021 Mar 7. No abstract available. PMID 33691182